CLINICAL TRIAL: NCT02386501
Title: A Phase 1b Dose Escalation Study of ADXS31-164 in Subjects With HER2 Expressing Solid Tumors
Brief Title: Dose Escalation Study of ADXS31-164 in Subjects With HER2 Expressing Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 164-05
Record Dates: First submitted 2015-02-26; First posted 2015-03-12 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: HER2 Expressing Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADXS31-164 (Experimental): Dose/Potency 5 x 108 CFU; 1 x 109 CFU; 5 x 109 CFU; 1 x 1010 CFU
  Interventions: Drug: ADXS31-164

INTERVENTIONS:
Drug: ADXS31-164

SUMMARY:
This is a Phase 1b, multicenter, open-label, dose-escalation study designed to estimate the maximum tolerated dose (MTD) and determine the recommended Phase 2 dose (RP2D) of ADXS31-164. Once the RP2D has been selected, up to 4 expansion cohorts will be evaluated.

DETAILED DESCRIPTION:
This is a Phase 1b, dose-escalation, open-label study in subjects with HER2 expressing solid tumors. Subjects will receive escalating doses of ADXS31-164 every 3 weeks during a 12-week treatment cycle. Subjects will receive a prophylactic regimen completed at least 30 minutes prior to each ADXS31-164 infusion to mitigate and manage the potential immune response seen with immunotherapy administration. In addition, all subjects will participate in a 3 year Lm surveillance period. The surveillance period will begin following the last dose of study treatment or at the time of study discontinuation. This period is intended to help ensure the eradication of Lm bacteria. This period will also include a 6- month course of trimethoprim/sulfamethoxazole which will be initiated approximately 72 hours after the completion of the last dose of ADXS31-164 or immediately following study discontinuation. In subjects with a sulfa allergy, the 6-month course should consist of ampicillin 500 mg 4 times daily initiated approximately 72 hours following the last dose of study treatment or immediately following study discontinuation.

Dose escalations and de-escalations will be dictated by a 3+3 design. Three dose levels may be evaluated during the dose escalation portion starting with Dose Level 1 at 1 x 109 colony forming units (CFU). Once the Maximum Tolerated Dose (MTD) and RP2D have been identified, up to 4 HER2 overexpressing tumor specific expansion cohorts will be evaluated. The specific tumor types included in the expansion cohorts may include breast and gastric cancer with the remaining to be determined by the sponsor after review of data from Part A. Treatment cycles can be repeated at the RP2D (or less) for each subject for up to 2 years, until a study discontinuation criterion is met or he/she has completed >6 months of study therapy and at least 1 cycle of treatment post observation of a complete response (CR)

ELIGIBILITY:
Inclusion Criteria:

* HER2 Positive
* Have histological or cytological diagnosis of locally advanced/metastatic HER2 solid tumors that has progressed or become intolerant to standard therapy or for which no standard therapy is available
* Have measurable and/or evaluable disease based on RECIST 1.1.
* ECOG performance status of 0 to 1

Exclusion Criteria:

* Is newly diagnosed with a curative treatment option available.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of' immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior monoclonal antibody therapy within 2 weeks prior to study Day 1. (Prior anti-HER2 therapy is acceptable).
* Has received anticancer chemotherapy, surgical treatment, and/or radiation therapy (except palliative radiation therapy for disease-related pain with a consult with the sponsor's medical monitor) within ≤2 weeks of first study treatment.
* Is dependent on, currently or has received within the past 4 weeks corticosteroids (hormone replacement therapy, topical corticosteroids and occasional inhaled corticosteroids are allowed).
* Has a contraindication to administration of trimethoprim/sulfamethoxazole or ampicillin.
* Has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)). NOTE: More common devices and prosthetics which include arterial and venous stents, dental and breast implants, and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any subject who has any other device and/or implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities for each dose level as assessed by CTCAE v 4.0 | 4 Months
Frequency and severity of adverse effects as assessed by CTCAE v 4.0 | 3 Years
  The type, incidence, severity, and causality of each AE, the duration of the event, and any required treatment interventions will be tabulated.

SECONDARY OUTCOMES:
Proportion of patients who have objective tumor response (complete or partial) | 3 Years
  Tumor response will be evaluated by RECIST 1.1 and irRECIST criteria.
Changes in clinical immunology based upon serum | Baseline through 12 Weeks
  Immunologic effects will be measured and evaluated by collection of peripheral blood for preparation of peripheral blood mononuclear cells (PBMCs) and serum at baseline, prior to each treatment and posttreatment in the first treatment cycle only.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Not Yet Recruiting, Los Angeles, California
  - Site, Aurora, Colorado
  - Grand Rapids, Michigan
  - Site, Charlotte, North Carolina
  - Site, Philadelphia, Pennsylvania
  - Dallas, Texas